CLINICAL TRIAL: NCT06976645
Title: Evaluation of the Upper Eyelid Dynamics in Simple Congenital Blepharoptosis Before and After Levator Muscle Resection Using High Speed Videography
Brief Title: Upper Eyelid Dynamics in Pediatric Blepharoptosis Using High Speed Videography
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Zamzam Mohamed Alham, Assistant lecturer, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UEL dynamics in cong.ptosis
Record Dates: First submitted 2025-04-03; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Upper Eyelid Dynamics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Levatot muscle resection (Other): Levator muscle resection for correction of upper eyelid congenital blepharoptosis
  Interventions: Procedure: Levator muscle resection

INTERVENTIONS:
Procedure: Levator muscle resection — Levator muscle resection

SUMMARY:
Evaluation of the Upper Eyelid Dynamics in Simple Congenital Blepharoptosis before and after Levator Muscle Resection Using High speed Photography

DETAILED DESCRIPTION:
Normal eyelid dynamics are essential for optimum performance and protection of the eye including distribution of the pre-corneal tear film, clearance of debris, stimulation of Meibomian gland secretion, and assistance of tear drainage via generating negative pressure in the lacrimal sac. Conversely, abnormal eyelid dynamics can have a variety of implications in ocular surface health and visual function.1 Current methods for evaluating eyelid dynamics include magnetic-based devices, high-speed videography, infrared videography, and direct observation.2-3 Whereas magnetic search coils are considered the gold standard for research purposes, they may not be practical at the clinical setting. Conversely, a readily available and cost-effective technology of smartphone video cameras with high speed video photography options has reached a level of perfection that may enable them to be used for objective and quantative slow motion analysis of eyelid dynamics.

The interest in the study of lid dynamics started early in 1977 through dynamic measurements made with a mechanical transducer connected physically to the upper eyelid. 4 The normal spontaneous blink rate has a wide variability, ranging from 2 to 50 blinks per minute. It is reported that normal blink duration varies from 300 to 572 milliseconds. Normal blink amplitudes also vary from 7.4 to 12.8 mm and decrease with age.5-6,7-8 Most of these values have been established with different techniques for analysis with magnetic search coil.6,7,9 High-speed cameras provide precise, measurable movement detection.9 With these cameras, the upper and lower eyelids have shown to both move also horizontally during the closure phase of eyelid blinking.7 Previous studies measured the spontaneous eyelid blink dynamic changes using a high-speed camera in various conditions as age-related changes5, following upper eyelid blepharoplasty and its association with dry eye10 and in patients with thyroid disease11.

Upper eyelid surgery can change the lid dynamics. For instance, incomplete lid closure is sometimes encountered after upper blepharoplasty. The most common cause of lagophthalmos is excessive skin resection, which acts as a negative passive force that is much stronger than the active closing force of the orbicularis oculi muscle and can disturb blinking .12 Congenital ptosis is the presence of an abnormally low position of the upper eyelid, with respect to the visual axis in the primary gaze .13 It may not be immediately noticeable after birth but is usually manifest within a few months. It can be unilateral or bilateral. It has a significant functional and psychosocial impact on the child.14The underlying etiology appears to be localized muscle dysgenesis. In the affected levator muscle fibers are infiltrated or replaced with fibrous and adipose tissue, which results in abnormal contraction and relaxation .15 There is an association between congenital ptosis and under action of the superior rectus muscle in up to 25% of unilateral cases and in 65% of bilateral cases .16 It may be associated with lagophthalmos on downgaze with exposure of the cornea. There is often a decreased or absent lid crease .13 Levator resection is the gold standard of surgical correction of simple congenital ptosis with fair to good levator function. It creates optimal lid contour and symmetry with relatively desirable cosmetic outcomes17-19. Lagophthalmos is one of the surgical consequences. It usually improves with time .20 In the study of Cruz et al.,2014 21 on supramaximal levator resection, spontaneous blinks were abnormal in 93% of the operated eyelids. The mean amplitude of the abnormal blinks was 37.1% of the contralateral eyelids. Downward eyelid saccades were reduced in 79% of the eyelids.

To the best of our knowledge this is the first study to assess the changes of eyelid dynamics in patients with simple congenital ptosis before and after levator muscle resection using high speed video photography. Aim of the study

Quantative subjective analysis of upper eyelid dynamics in patients with simple congenital ptosis before and after levator muscle resection using high speed video recording.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed as simple congenital ptosis with fair to good levator function (≥5 mm lid elevation) with age range from 5 to 18 years old.

Exclusion Criteria:

* Patients with a history of previous eyelid surgery or trauma

  * Blepharophamosis and Marcus Gun Jaw-winking syndrome
  * Patients with associated neurological disorders
  * Patients with craniofacial abnormalities
  * Patients with suspected myasthenia or myopathies
  * Patients with absent Bell's phenomenon
  * Patients with dry eye
  * Uncooperative patients

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Determine the changes of blinking velocity before and after levator resection in patients with congenital ptosis | One year
  Record the changes of blinking velocity in patients with congenital ptosis before and after levator resection &normal patients in same age group using high speed videography to detect changes in blinking velocity .

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mohamed Elshafei, Professor, Study Director — Minia University

REFERENCES:
- [Background] Hung G, Hsu F, Stark L. Dynamics of the human eyeblink. Am J Optom Physiol Opt. 1977 Oct;54(10):678-90. doi: 10.1097/00006324-197710000-00005. PMID 605924
- [Background] DeAngelis KD, Rider A, Potter W, Jensen J, Fowler BT, Fleming JC. Eyelid Spontaneous Blink Analysis and Age-Related Changes Through High-Speed Imaging. Ophthalmic Plast Reconstr Surg. 2019 Sep/Oct;35(5):487-490. doi: 10.1097/IOP.0000000000001349. PMID 30844914
- [Background] Mak FHW, Ting M, Edmunds MR, Harker A, Edirisinghe M, Duggineni S, Murta F, Ezra DG. Videographic Analysis of Blink Dynamics following Upper Eyelid Blepharoplasty and Its Association with Dry Eye. Plast Reconstr Surg Glob Open. 2020 Jul 21;8(7):e2991. doi: 10.1097/GOX.0000000000002991. eCollection 2020 Jul. PMID 32802679
- [Background] Wuthisiri W, Peou C, Lekskul A, Chokthaweesak W. Maximal Levator Resection Beyond Whitnall's Ligament in Severe Simple Congenital Ptosis with Poor Levator Function. Clin Ophthalmol. 2022 Feb 17;16:441-452. doi: 10.2147/OPTH.S340781. eCollection 2022. PMID 35210749
- [Background] Allard FD, Durairaj VD. Current techniques in surgical correction of congenital ptosis. Middle East Afr J Ophthalmol. 2010 Apr;17(2):129-33. doi: 10.4103/0974-9233.63073. PMID 20616918